CLINICAL TRIAL: NCT02642172
Title: A Randomized, Double - Blind Study With Two Parallel Arms for 4 Months (20 Weeks), Evaluating the Effectiveness of the Prebiotics in Patients With Non-alcoholic Liver Disease.
Brief Title: Prebiotics in Patients With Non-alcoholic Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaplan Medical Center (Other)
Responsible Party: Principal Investigator, Yaakov Maor, Principal Investigator, Kaplan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PN-837-CTIL
Record Dates: First submitted 2015-12-13; First posted 2015-12-30 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Non-alcoholic Fatty Liver Disease; Metabolic Syndrome
Keywords: Inulin, OFS (oligofructose)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Metabolic Syndrome | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ITF (Inulin/OFS 75/25) (Experimental): 16 gram/day of ITF (Inulin/OFS 75/25)
  Interventions: Dietary Supplement: ITF (Inulin/OFS 75/25)
- placebo (Placebo Comparator): 16 gram/day of maltodextrin (placebo)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: ITF (Inulin/OFS 75/25) — Participants will consume 16 g/day ITF
  Other Names: Prebiotics- Inulin, OFS - oligofructose
  Arms: ITF (Inulin/OFS 75/25)
Dietary Supplement: Placebo — Participants will consume 16 g/day maltodextrin
  Other Names: maltodextrin
  Arms: placebo

SUMMARY:
The purpose of this present study is to evaluating whether prebiotics - ITF (Inulin/OFS 75/25) is effective in treating patients with non-alcoholic liver disease.

DETAILED DESCRIPTION:
The study will include 60 patients with Non-alcoholic fatty liver disease (NAFLD) which will randomize to two groups, receiving either ITF (Inulin/oligofructose-OFS 75/25) or maltodextrin (placebo).

The trial will last for 26 weeks: Stage 1-Run-in period: Subjects will be followed to ascertain weight maintenance. Stage 2- Randomized intervention period: Subjects will be assigned to receive 16 gram/day of ITF or maltodextrin. Both ITF and placebo will be provided in identical opaque packages and both subjects and researchers will be blinded to the content.

After signing informed (-2 week) consent, the following data will be collected: demographics, lifestyle habits including dietary questionnaires, and medical history. At week 0, week 12 and week 24 all the following tests will be performed: Vital Signs: blood pressure, anthropometric measurements, body composition determined by bioelectrical impedance analysis (BIA). Biochemical blood tests: liver function tests fasting glucose insulin & lipid profile, CRP (an inflammation marker), SCFA, BCAA, and LBP and FGF 19. Fecal samples: fecal samples will be used for microbiota composition analysis, and BA analysis. Assessment of liver status At week 0 and 24 by using magnetic resonance spectroscopy (1H-MRS), SteatoTest and NashTest (FibroMax™) and by liver enzymes for evaluating steohepatitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NAFLD based on fatty infiltration detection by ultrasonography and alanine aminotransferase levels of (ALT) ≥ 30 U/L male ≥ 19 U/L females.
* Over-weight (BMI ≥ 27 kg/m2) who fulfill the criteria of the National Cholesterol Education Program (NCEP) metabolic syndrome
* Willing to sign informed consent to participate in the study
* Patients without diabetes or with well-controlled diabetes (HbA1C < 7.5%) who are treated by diet ± metformin

Exclusion Criteria:

* Pregnancy
* Uncontrolled diabetes
* Diabetic treatment other than metformin, unusual diets (vegetarian, vegan), usage of antibiotics, probiotics or prebiotics up to 6 months prior to study, alcohol abuse, presence of gastrointestinal or mental disorders, weight-loss treatment, bariatric surgery
* Serious medical conditions
* Evidence of another etiology for chronic liver disease such as: hepatitis B, hepatitis C, HIV, autoimmune diseases and metabolic diseases, medications with known hepatotoxicity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the severity of NAFLD | 12 weeks
  Determined by
  1. liver fat fraction measured by magnetic resonance spectroscopy (1H-MRS)
  2. Blood test for calculate Inflammation score using SteatoTest and NashTest (FibroMax™)
  3. Blood test for liver enzyme

SECONDARY OUTCOMES:
Change from baseline of gut microbiota composition. | 12 weeks
  Quantitative evaluation of the change in the composition of bacteria from stool samples
Change from baseline in glycemic control | 12 weeks
  Determine by OGTT.
Change from baseline in insulin sensitivity | 12 weeks
  Which will be determined by a fasting Glucose and Insulin blood tests and Calculate homeostasis model assessment (HOMA).
Change from baseline in lipid profile | 12 weeks
  Which will be determined by blood test for lipid profile - Triglycerides, cholesterol-LDL and cholesterol-HDL

CONTACTS AND LOCATIONS:
Overall Officials: Yaakov Maor, Dr, Principal Investigator — Kaplan Medical Center
Locations (1):
- Kaplan Medical Center, Rehovot, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dewulf EM, Cani PD, Claus SP, Fuentes S, Puylaert PG, Neyrinck AM, Bindels LB, de Vos WM, Gibson GR, Thissen JP, Delzenne NM. Insight into the prebiotic concept: lessons from an exploratory, double blind intervention study with inulin-type fructans in obese women. Gut. 2013 Aug;62(8):1112-21. doi: 10.1136/gutjnl-2012-303304. Epub 2012 Nov 7. PMID 23135760